CLINICAL TRIAL: NCT01329107
Title: Efficacy of a Multimodal Rehabilitation Program to Bladder Cancer Patients
Brief Title: Multimodal Rehabilitation Program to Bladder Cancer Patients
Acronym: MRPBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M20100122; Aarhus University (Other Grant/Funding Number: Aarhus University)
Record Dates: First submitted 2011-03-10; First posted 2011-04-05 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Bladder Cancer
Keywords: Rehabilitation; Enhanced Recovery; Health related Qouality of Life; Patient outcomes
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention): Standard Care
- Multimodal intervention (Experimental): Intervention group will be assigned to specific decribed multimodal intervention
  Interventions: Behavioral: Multimodal Intervention

INTERVENTIONS:
Behavioral: Multimodal Intervention — Patients in the intervention group will be taught to manage their new urinary diversion BEFORE operation. Traing kit will be provided so they can train the procedure forehanded. Second they will get a personally physical training program to optimize the total body function before operation. Nutritional status will be meassured and appropriate advices will be given BEFORE operation.
  After operation the intervention group will be mobilised in a fast speed compared to standard care.
  Other Names: Enhanced care programme; Fasttrack pathways
  Arms: Multimodal intervention

SUMMARY:
The incidence of bladder cancer is increasing. Denmark have approximately 1800 incidence per year. The disease is most frequently in males above the age of 70 years. In invasive bladdercancer surgery including removal of the seak bladder with constructing of a new diversion, is the first line treatment. However the procedure is followed by a high morbidity and convalescence. Extended surgical procedure cause pain, stress-induced metabolism and impaired organ function resulting in postoperative complications impacting on rehabilitation. The combination of extended surgery and the increasing numbers of elderly comorbid patients with invasive bladder cancer challenge professional treatment and care

The aim of the study is to investigate the efficacy of a multiprofessional rehabilitation programme for patients with invasive bladder cancer referred to surgery

Material and Methods The study is a randomised controlled trial. All patients > 18 years referred to radical cystectomy will be eligible for this study. The efficacy is primary expressed by the difference in length of stay(LOS). Secondly by complications, health related quality of life(HRQoL) and patient reported quality of care during hospitalization. The intervention includes precise instructions and educations in intensive pre- and postoperatively exercises and stoma-care, supported by the multiprofessional team.

Perspective It is a national goal to improve cancer care. This study is of critical importance and places great emphasis on the patients perspective and involvement in a successful outcome for participant's and involvement in nutritional support, intensive exercises and stoma care, supported by the multidisciplinary team

DETAILED DESCRIPTION:
PhD protocol

Efficacy of Multi-professional Rehabilitation in Patients with Bladder Cancer (offered radical cystectomy)

Bente Thoft Jensen, RN, MPH, research nurse Department of Urology Aarhus University Hospital, Skejby

Supervisors:

Michael Borre, associate professor, DMSc, PhD, Department of Urology, Aarhus University Hosptial, Skejby (head supervisor).

Klaus Ernst-Møller Jensen, consultant, DMSc, Department of Urology, Aarhus University Hospital, Skejby

Sussie Laustsen, associate professor, PhD, Clinical Institut, Aarhus University

Mette Krintel Petersen, post-doc, PhD, research physiotherapist, Department of Physiotherapy and Occupational Therapy, Aarhus University Hospital, Skejby

Collaborators:

Department of Physiotherapy and Occupational Therapy, Aarhus University Hospital, Skejby Mette Borre, dietician, Department of Gastroenterology and Hepatology, Aarhus University Hospital, Aarhus Sygehus, Norrebrogade Berit Kiesby, stoma-care nurse, Department of Urology, Aarhus University Hospital, Skejby

Background In Denmark, the incidence of patients with bladder cancer is approximately 1800 cases annually; 75% of the cases are men. The disease is most frequent among the 50 to 80-year-olds and most cases are approximately 70 years old [1]. Recent studies have shown that the incidence of bladder cancer is increasing in Europe[2]. Cystectomy is one of the most comprehensive surgical procedures in urology[3,4]. In Denmark, the average post-operative length of stay (LOS) was 19 days in 2005; the hospital mortality rate was 3.7% and 58% had a complicated course of disease. The mortality was comparable to experiences abroad [3,5]. LOS is, however, long compared with high-volume hospitals with well-defined clinical patient pathways [1,5,6]. Major surgery causes pain and stress-induced catabolism leading to an unwanted metabolic and inflammatory response, impaired organ function and risk of thrombosis. These conditions increase the risk of losing muscle mass and reduce the activity level [2]. Overall, the above-mentioned circumstances delay the rehabilitation process. The concept "fast-track surgery" is a multi-modal and inter-professional approach to reduce post-surgical morbidity and optimise post-surgical rehabilitation [7,8].

The multi-modal approach comprises both pre-operative optimisation of organ function, patient education, effective pain management, early post-operative mobilisation and early oral nutrition [9]. The concept has proven effective, though primarily documented in connection with colorectal surgery [9-11,12,13,], with increased survival, reduced LOS and reduced costs compared with conventional patient pathways[14,15]. The combination of a major surgical intervention and an increasing number of elderly comorbid patients with bladder cancer poses a challenge to treatment and care in all phases of the patient pathway. The above studies primarily focus on the pre- and post-operative effort. Evidence is sparse concerning the importance of an optimised pre-operative effort in rehabilitation [11]. It is hypothesised that an optimised patient pathway calls for an inter-professional pre-operative clinical evaluation and a pre-optimisation of the patient's general condition including nutrition and physical activity[11,16-18]. There is low evidence of the efficacy of multi-modal pre-optimisation efforts in major surgical procedures in urology [2,19]. Especially concerning the importance of a multi-facilitated pre-operative intervention for rehabilitation and health-related quality of life [7,8]. Generally, there has been a post-operative effect concerning early nutritional intervention and LOS [20]. Early nutritional intervention increases the number of patients fulfilling the threshold for sufficient nutritional status [15,21]. Nutrition strategies are increasingly combined with physical training consisting of exercise to increase muscle strength and endurance, to increase hypertrophy of muscle cells by increasing muscle protein synthesis and reducing disintegration [22]. Thus, a pre-operative multi-modal intervention involving nutritional optimisation and physical training should be a part of future studies. A muli-modal patient pathway will involve expectations of an increased risk that the economic burden will shift to the primary sector [23], an increased frequency of readmissions, complications and reduced quality of life. This thesis investigates the efficacy of pre- and post-operative multi-modal interventions in the rehabilitation of patients with bladder cancer undergoing cystectomy.

Material: All patients undergoing cystectomy at Aarhus University Hospital in 2009 fulfilling the inclusion criteria.

Study A. To investigate the efficacy of pre- and post-operative multi-modal intervention in bladder cancer patients referred to radical cystectomy

The following hypotheses are tested:

* An inter-professional multi-modal pre- and post-operative intervention promotes rehabilitation and reduces length of stay
* The intervention group obtains a higher functional and activity level compared with the control group
* The intervention group obtains a better management of urinary diversion compared with the control group

Material and methods:

Primary endpoints: LOS is defined as number of post-operative days (until 7 defined discharge criteria are fulfilled). The outcome data will be presented approximately 12 months after inclusion have been closed

Secondary endpoints:

* complications ( measured at discharge and 120 days postoperatively in average)
* Activity and functional level( will be measured every day during admission and 120 days after discharge).Pfysical parametres like bioimpedance, musclepower and handgrip strength will be measured at baseline( two weeks before operation, one day before operation, at discharge and 120 days after operation in both arms)
* Patient-experienced quality during admission ( measured with EORTC-questionaire at discharge in both arms)Informations will be presented approximately 12 months after inclusion is closed
* Health-related quality of life will be measured at baseline and 120 days after operation ( EORTC questionaire).
* Management of urinary diversion will be measured at baseline, before operation,35 days and 120 days after operation.A validated stoma score scale for patient stoma skills will be used.The outcome data will be presented approximately 12 months after inclusion have been closed

Sample size. The study population is calculated on the basis on LOS for patients undergoing cystectomy at the Department of Urology, Aarhus University Hospital, Skejby in 2008. Average LOS was 13 days with a standard deviation of 4.75 days. Risk of type 1 error was 5% at a 2-sided analysis and strength at 80%. Lowest relevant difference in effect is a 20% reduction in LOS in the intervention group. When a 2-sided comparison is made, 92 patients have to be included; 46 in the intervention and control group, respectively.Written information about the study is forwarded to the patients along with the appointment for a uro-oncological evaluation.

Randomisation: Performed 14-17 days prior to surgery. When deciding on surgery the patient receives oral information about the examination. After time for deliberation and giving informed consent, the patients are randomised at the outpatient consultation following the uro-oncological evaluation.

Monitoring:

Demographic and clinical background variables are registered at baseline. Follow-up after 4 months. Data are collected for further analysis at 1-year follow-up (appendix 1.1-1.5). All patients undergo nutritional screening at baseline by NRS [32,33].

Patients with age-adjusted score<3 will receive supplements according to standard criteria[25-28]. Energy demand is calculated as weight x100x1.3 KJ /day. Protein need is calculated as weight x 1.5 gram protein/day. Fluid need is calculated as weight x 30 ml/day [30]. Comorbidity is scored using the Charlson index score, pain and nausea using the VAS-score [32,33].Habitual intestinal function is scored using the Bristol scale[34].

Physical activity level is estimated at baseline using the Physical Activity Scale (PAS) [35]. Daily mobilisation time and walking distance are registered pre-operatively and during admission using a pedometer [36,37].

Ability to perform personal activities of daily living are evaluated daily during admission using the KATZ score [38].

Muscle power, muscle strength and body composition are registered at baseline, pre-operatively, at discharge and 35, 120 (and 365) days post-operatively. Muscle power (force x velocity) is evaluated by leg extensor power Rig [39]; Isometric muscle strength (hand grip strength) is evaluated by "Good Muscle Strength" [40]and body composition is evaluated by bioimpedance [41] Progression in management of urinary diversion is evaluated by a categorial scale (appendix 1.4).

Standard treatment:

Patients eat normally until the operation. The rectal ampulla is emptied the evening before surgery. From midnight the patients fast and drink two glasses of sweet juice at 06.00 am before the operation. TED stockings are used to prevent thrombosis per- and post-operatively until the mobilisation criteria have been met. 5000 IU of Fragmin are injected subcutaneously from day 0. Individual prescriptions are made for patients with sclerotic diseases. Per-operative infection prophylaxis is standardised.

Sevofluorane is used as a sedative and Bupivacain as well as Ultiva infusions as pain management. Epidural catheter is used for pain treatment at th-12-L1 level. The transfusion regime is standardised. Pain treatment: Post-operatively - epidurally administered Bupivacain 2.5 mg /ml 5-6 ml / h in 3 full days. Peripheral pain treatment is tablet paracetamol 1g x 4 and from day 2, two tablets Ibuprofen 400 mg x 3.

* Care of urinary diversion; When surgery is decided there is an interprofessional meeting concerning management of stoma and neobladder. Stoma markings are made the day before surgery in collaboration with the surgeon, the patient and the stoma care nurse. Relevant aids are demonstrated and the post-operative regime is presented.
* Physiotherapy: Instruction and information about pulmonary physiotherapy is performed pre-operatively. Daily mobilisation in each shift post-operatively.
* Discharge criteria (see appendix 1.5)

Intervention

In addition, the following initiatives are made in the intervention group:

* Pre-operative optimisation: The intervention group is taught pre-operatively about the management of urinary diversion. Exercise kit is handed out with exercises to perform in the home. Intensive instruction and teaching is provided by physiotherapist. Moreover, plans for post-operative progressive mobilisation and transfer techniques. Balancing mutual expectations for the entire intervention.
* Post-operative optimisation: Intensive, structured and progressive plans for daily mobilisation and physical activity from the day of surgery until planned discharge at 7-9 post-operative day as well as instruction in urinary diversion by the stoma care nurse.

Effect: Expressed as the difference in: LOS, complications, functional and activity level and management of urinary diversion.

Statistics: Normally distributed data are described as mean, standard deviation (SD) and 95% confidence intervals (CI) and tested with Student's t-test for paired data, unpaired data are tested by unpaired t-test and repeated measurements. Non-normally distributed data are described as median and range and tested by the Mann-Whitnew U-test or Wilcoxon's sign rank test. When testing 3 or more variables the Friedman test is applied. Pearson's test is applied in correlation analyses if conditions are met or Spearman's Rho. Frequencies are compared by Fischer's exact test. Associations between variables are reported as odds ratios and 95% CI.

Study B: Health-related quality of life and experienced patient quality in multi-modal interventions

Purpose: to study the effect of multi-modal interventions concerning the patient experience during hospital admission and health-related quality of life (HeQoL).

Hypothesis:

The intervention group will have better experienced quality and higher HeQoL. End points: Score concerning HeQoL and patient experienced quality. Material /Method: Same method and study population as in study 2. Disease-specific questionnaires from the European Organisation for Research and Treatment of Cancer, EORTC QLQ-BLM30 and QLQ-C30 [42] were applied. Scores are made at baseline and follow-up at planned control visits (35 days, 120 days and 365 days). At discharge EORTC In-PATSAT32 is used to evaluate the patient experience of quality during admission. All questionnaires are validated and translated into Danish [43,44].

Statistics study B. Data are registered at a categorial scale and described as mentioned in study A for non-normally distributed data. Wilcoxon's sign rank test is used to test the difference in HeQoL between the groups.When testing 3 or more groups, Friedman's test is applied. Spearman's Rho is used for correlation analyses of non-normally distributed data. Associations between variables are reported as ORs and 95% CI.

Ethical considerations: The study is approved by the Central Denmark Committee on Biomedical and Research Ethics and the Danish Data Agency. Transport costs in connection with control visits are refunded and it is attempted that examinations take place at days where the patient has to meet for a control visit at the hospital. At present, the treatment offer to this patient group does not include pre- and post-operative optimisation and it is not deemed unethical to randomise patients to pre- or post-operative optimisation or standard treatment, respectively. The study is registered in the American clinical database www.clinicaltrials.gov.

Research plan including time schedule: Daily project management, data processing and statistical analyses will be made and interpreted by PhD student Bente Thoft Jensen(BTJ), who is also responsible for publication of results. Data collection will be made in collaboration with the stoma care and nutrition responsible nurses and a dietician. Instruction in home exercises, test of functional and activity level is made in collaboration with the physiotherapists in the bladder team. The project is expected to start in the spring 2011. Inclusion of patients will run for 1.5 years according to the current surgical activity. Data collection and analyses are made in 2011 and 2012. Summary and reporting of results will be made in 2012.

Publication: The project results are communicated in 3 peer-reviewed articles and in a PhD thesis.

Funding:The project will be partly financed by the Department of Urology, Aarhus University Hospital, Skejby (1/3), by the hospital management teat, Aarhus University Hospital, Skejby (1/3) and the rest will be university scholar ships, industrial collaborators and foundations.

Perspective: Cystectomy is one of the most resource-consuming surgical procedures. Despite comprehensive shifts in paradigms in both nursing and treatment strategies throughout the last decade, the average LOS has only been modestly reduced. In addition to the newly introduced packages for diagnostics and treatment of cancer patients it is essential to strengthen the overall effort. This PhD project should be seen as a part of the endavour to fulfil all parts of the overall purpose concerning evidence-based optimisation of the rehabilitation of bladder cancer patients. Whether urological patient pathways with a pre-operative intervention can minimise post-operative complications, lead to a higher HeQoL and shorten the rehabilitation period will be highlighted.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years referred to radical cystectomy at the Department of Urology, Aarhus University Hospital, Skejby because of invasive bladder cancer.

* Must have accepted the operation procedure
* Must have accepted the pre and post-operative careprogram
* Patients must be able to read and write in Danish.

Exclusion Criteria:

* patients with neuro-muscular and cognitive diseases
* Patients referred because of voidingdysfunctions
* Patients with general bad condition ( judged by the surgeons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of a Multimodal Rehabilitation Program to Bladder Cancer Patients | 2 yrs. Due to the rate of operation pr week the inclusion will close in the beginning of 2013
  * Primary Endpoint is the difference in the length of stay (LOS) between the standard care gruop and the intervention group.
  * LOS will be measuared when the 7 defined standard discharge criteria are fulfilled. The difference between the primary outcome will be compared and published approximately 12 months after inclusion is closed

SECONDARY OUTCOMES:
Efficacy of Multimodal Rehabilitation Program to Bladder Cancer Patients | 2yrs. Due to the rate of operations pr week the inclusion will close in the beginning of 2013
  * HeQoL will be measured at baseline and 120 days postoperatively.( EORTC questionaire)
  * Complications postoperatively will be meassured at discharge and at 120 days postoperatively with the listed domaines on the Memorial Sloan Kettering Tool.
  * Management of the urinary diversion will be measured on a patient stoma skill score ( baseline, before operation, +35 days and at 120 days)
  * All outcomes is expected to be published in 12 months on average after operation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borre, PH.D, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Michael Borre, Aarhus, Aarhus N
  - Aarhus University Hospital, Aarhus